CLINICAL TRIAL: NCT06867861
Title: Effect of Fiber Supplementation on the Need for Medication With Gestational Diabetes: A Randomized Controlled Trial
Brief Title: Effect of Fiber Supplementation on the Need for Medication With Gestational Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Jerri Waller, Principal Investigator, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-08-FB-0214
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational Diabetes Mellitus; Fiber; GDM
MeSH Terms: conditions — Diabetes, Gestational | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fiber (Experimental): Participants will psyllium fiber supplement capsules, 2g soluble fiber per capsule. They will be instructed to take 4 capsules twice daily for a total of 16g supplemental soluble fiber per day. This will be continued throughout pregnancy.
  Interventions: Dietary Supplement: Fiber
- No Fiber (No Intervention): Participants will receive no fiber supplementation capsules.

INTERVENTIONS:
Dietary Supplement: Fiber — Psyllium fiber supplement capsules, 2g soluble fiber per capsule. They will be instructed to take 4 capsules twice daily for a total of 16g supplemental soluble fiber per day. This will be continued throughout pregnancy.
  Arms: Fiber

SUMMARY:
The hypotheses to be tested are 1) Fiber supplementation will decrease the need for medication in patients with gestational diabetes, and 2) Fiber supplementation will decrease adverse maternal and neonatal outcomes in these patients. In this study, the investigators will conduct a randomized controlled trial to limit bias in evaluating these hypotheses.

DETAILED DESCRIPTION:
The study team proposes a randomized controlled trial of women with singleton pregnancies who present with a new diagnosis of diet-controlled gestational diabetes (previously referred to as GDMA1). The participants will be randomized to the intervention group (fiber supplementation) or control group (no fiber supplementation) in 1:1 fashion. The participant will be randomized by a number-generating computer software after recruitment at the new gestational diabetes education class.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Known or new diagnosis of gestational diabetes without reason for medication
* Age >=18 to <=50

Exclusion Criteria:

* - Non-English as primary language.
* Known or suspected fetal anomaly or aneuploidy.
* Known lower bowel disorder
* Known phenylketonuria
* Prisoners.
* Management of diabetes outside of Eastern Virginia Medical School Maternal Fetal Medicine.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Need for GDM Medication | From date of randomization until the date of first documented progression (assessed up to 7 months)
  The primary outcome is the need for medication (either insulin or oral hypoglycemic agents) for management of gestational diabetes (progression from GDMA1 to GDMA2). We chose this primary outcome because the need for medication is associated with the need for significantly more antenatal interventions due to increased adverse pregnancy outcomes.

SECONDARY OUTCOMES:
Hgb A1c at delivery | At delivery
  Measurement of Hgb A1c
Rate of Fetal Demise | From date of randomization until the date of documented occurrence (assessed up to 7 months)
  Rate of fetal demise
Number of Participants Diagnosed with Fetal Growth Restriction | From date of randomization until the date of first documented progression (assessed up to 7 months)
  Number of participants diagnosed with fetal growth restriction
Number of Participants Diagnosed with Preeclampsia | From date of randomization until the date of first documented progression (assessed up to 7 months)
  Number of participants diagnosed with preeclampsia
Number of Participants with Placental Abruption | From date of randomization until the date of first documented progression (assessed up to 7 months)
  Number of participants with placental abruption
Mode of Delivery | At delivery
  Rates of cesarean and vaginal deliveries
Indication for Cesarean Delivery | At delivery
  Rates of each indication for cesarean delivery
Rate of Shoulder Dystocia | At delivery
  Rate of shoulder dystocia
Quantitative Blood Loss | At delivery
  Blood loss in mL
Rate of Postpartum Hemorrhage | At delivery
  Rates of patients with quantitative blood loss > 1000mL
Rates of Infection | Delivery until discharge (assessed up to 5 days)
  Rates of infection
Birth Weight | At delivery
  Birth weight
Apgar Score | At delivery
  Apgar scores at delivery on a scale of 0 to 10, with higher scores meaning a better outcome
Rates of Neonatal Infections | Delivery until discharge (assessed up to 5 days)
  Rates of neonatal infections
Rate of Respiratory Distress Syndrome | At delivery
  Rate of respiratory distress syndrome
Rate of Necrotizing Enterocolitis | Delivery until discharge (assessed up to 5 days)
  Rate of necrotizing enterocolitis
Rate of NICU Admission | Delivery until discharge (assessed up to 5 days)
  Rate of admission to NICU
Days in NICU | Delivery until discharge of the neonate (assessed up to 180 days)
  Days spent in NICU

CONTACTS AND LOCATIONS:
Overall Officials: Jerri Waller, MD, Principal Investigator — Macon & Joan Brock Virginia Health Sciences at Old Dominion University
Locations (1):
- Macon & Joan Brock Virginia Health Sciences at ODU, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, et al. A multicenter, randomized trial of treatment for mild gestational diabetes. Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. N Engl J Med 2009;361:1139-48.
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Karter AJ, Subramanian U, Saha C, Crosson JC, Parker MM, Swain BE, Moffet HH, Marrero DG. Barriers to insulin initiation: the translating research into action for diabetes insulin starts project. Diabetes Care. 2010 Apr;33(4):733-5. doi: 10.2337/dc09-1184. Epub 2010 Jan 19. PMID 20086256
- [Background] Chandalia M, Garg A, Lutjohann D, von Bergmann K, Grundy SM, Brinkley LJ. Beneficial effects of high dietary fiber intake in patients with type 2 diabetes mellitus. N Engl J Med. 2000 May 11;342(19):1392-8. doi: 10.1056/NEJM200005113421903. PMID 10805824
- [Background] Anderson JW, Allgood LD, Turner J, Oeltgen PR, Daggy BP. Effects of psyllium on glucose and serum lipid responses in men with type 2 diabetes and hypercholesterolemia. Am J Clin Nutr. 1999 Oct;70(4):466-73. doi: 10.1093/ajcn/70.4.466. PMID 10500014
- [Background] Sun J, Wang J, Ma W, Miao M, Sun G. Effects of Additional Dietary Fiber Supplements on Pregnant Women with Gestational Diabetes: A Systematic Review and Meta-Analysis of Randomized Controlled Studies. Nutrients. 2022 Nov 2;14(21):4626. doi: 10.3390/nu14214626. PMID 36364883
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574